CLINICAL TRIAL: NCT05118191
Title: Efficacy of Commercially Available Technology in Augmenting Sleep and Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Victor Finomore, Director of Applied Research, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2106353559
Record Dates: First submitted 2021-10-29; First posted 2021-11-11 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Sleep Quality
Keywords: Sleep; Commercial devices
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants will undergo 4 weeks of baseline data collection followed by 4 weeks of data collection while utilizing an assigned sleep augmentation device each night during sleep. Augmentation devices will be assigned with respect to 1) eligibility of inclusion/exclusion criteria of each device and 2) interest in participating with the available devices based upon responses in the qualifying survey on sleep preferences. If participants indicated that they were willing to try both the OOLER & the Embr Wave, & were eligible to do so, they will be randomly assigned a device based upon current availability. Women who experience menstrual flow will be scheduled to ensure that flow occurs on weeks 4 & 8 for consistency.
  Participants will complete daily, weekly, & monthly surveys, as well as weekly & monthly cognitive assessments. Participants will also have their sleep monitored nightly via the OURA ring & EEG headband. An additional exit survey will be completed at the end of week 8.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OOLER (Active Comparator): Participants will use the OOLER device.
  Interventions: Other: OOLER
- EmbrWave (Active Comparator): Participants will use the Embr Wave 2 device.
  Interventions: Other: EmbrWave

INTERVENTIONS:
Other: OOLER — Following the baseline block (first four weeks), participants will use the OOLER device to power a cooling mattress pad each night during sleep for four weeks.
  Arms: OOLER
Other: EmbrWave — Following the baseline block (first four weeks), participants will use the Embr Wave 2 device to provide pulsed warm sensations to the inner wrist each night during sleep for four weeks.
  Arms: EmbrWave

SUMMARY:
The objective of this research study is to assess how the implementation of various commercially available devices affect sleep quality, sleep structure, nocturnal physiology, subjective wellness, recovery from stressors, and resultant effects on performance and well-being.

DETAILED DESCRIPTION:
Sleep is a vital process for memory, cognitive performance, physical recovery, hormonal balance, and the repair of cellular damage, among numerous other functions. Despite its importance for maintaining one's health, it is amongst the most variable human behaviors experienced across the population. While many individuals fail to allocate sufficient time in their schedules for sufficient sleep, many individuals allocate plenty of time but struggle to receive efficient, and good quality sleep. In both cases, failure of the body to receive its required combination of enough and efficient enough sleep can result in significant consequences, including increased rates of disease development.

In an effort to help with these issues, which affect a significant portion of the adult population, commercial companies have sought to combine science, convenience, and good hygienic practices in the development of products aimed toward augmenting sleep. A wide range of products have hit the market including supplements (i.e. melatonin, melatonin infused products, GABA), sound producing devices (i.e. white noise machines), wearable products (i.e. sleep masks, special pajamas), and physiological modification devices and routines (i.e. temperature modulators, meditation), among dozens of other products, all with varying degrees of validity and scientific backing. Thermoregulatory products, the types of technologies utilized herein, have a great deal of scientific backing in how they have the potential to enhance sleep behaviors. Given the critical reduction in core body temperature that is needed at sleep onset, careful modulation of reduced body temperature is vital for falling asleep, staying asleep, and receiving good quality sleep. While these products demonstrate promising potential, further research is needed to identify the efficacy of these products in enhancing sleep. Further, it is of high interest what aspects of sleep can be enhanced via thermoregulation, what factors contribute to the degree of intervention impact, and what subsequent facets of overall well-being and performance are most improved by this type of sleep modulation.

ELIGIBILITY:
Inclusion Criteria:

• Male or female 18-50 years of age

Exclusion Criteria:

* Has a head diameter outside the range of 20.8-24 inches, or an approved head mounted EEG device doesn't otherwise fit properly
* Participants home is not air conditioned (exclusion for the OOLER only)
* Is pregnant or actively trying to become pregnant
* Has a known or diagnosed sleep disorder
* Females who have become menopausal or are exhibiting signs or symptoms of becoming perimenopausal
* Females who are unable to identify when their monthly menstrual period will occur
* Individuals who work during the night shift or have significantly abnormal sleep schedule
* Has undergone travel across more than two collective time zones in the last two weeks
* Individuals who intend to have any significant medical procedures scheduled to occur within 12 weeks of enrollment
* Individuals who have intentions, or have discussed with their doctor, about adding or making any alterations to their prescribed medications within 12 weeks of enrollment
* Individuals who have any travel plans or other obligations within 12 weeks of enrollment that would prevent them from completing study requirements and attending required laboratory visits
* Individuals who intend to make significant alterations to their sleeping patterns within 12 weeks of enrollment. This may include, but is not limited to, changes such as moving, getting a new mattress, having someone move in with them, etc.
* Does not meet the ACSM's guidelines for exercise prescription. This is defined as:

  1. Presenting with an absolute contraindication OR

     1. Has a known cardiovascular, pulmonary, renal, metabolic disease, or other chronic illness
     2. Presents with symptoms indicating cardiovascular, pulmonary, renal, or metabolic disease
  2. Presenting with two or more relative contraindications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Nocturnal Heart Rate as measured by OURA Ring | Daily from baseline through study completion at 8 weeks
  Heart rate (beats per minute) will be quantified throughout the night via the OURA ring.
Change in Subjective Sleep Quality measured via Questionnaire | Daily from baseline through study completion at 8 weeks
  A custom daily morning questionnaire will be used to record how a participant feels the quality of their sleep was the previous night (e.g. 1, very poor; 10 excellent). This questionnaire will be taken on the participants smartphone within 30 minutes of waking.
Change in Nocturnal Heart Rate Variability as measured by OURA Ring | Daily from baseline through study completion at 8 weeks
  Heart rate variability will be quantified throughout the night via the OURA ring.
Change in Eriksen Flanker Task | Changes from baseline versus end of study week 8
  The Flanker Task is a response inhibition test used to assess the participant's ability to suppress a response that is inappropriate based on the task rules. Participants are to respond, left or right, to the direction of the middle arrow (target arrow) of five aligned items. The task consists of congruent stimulus (the direction of the target arrow and flanker arrows are the same), incongruent stimulus (the direction of the target arrow is opposite of the flanker arrows), and neutral stimulus (flanker items are different then the target arrow). The dependent variable is the measurement of reaction time to select the direction of the target arrow.
Change in Psychomotor Vigilance Task | Changes from baseline versus end of study week 8
  A reaction time test that measures a person's sustained attention to a cue presented on a screen at random inter-stimulus intervals. In addition to the measures of reaction time to correct responses the errors of commission (responding when there is not response cue) and omission (failing to respond to a response cue).

SECONDARY OUTCOMES:
Change in Subjective Epworth Sleepiness Scale measured via Questionnaire | Weekly throughout study completion at 8 weeks
  Participants will complete previously validated questionnaires as often as weekly.
  Epworth Sleepiness Scale (ESS) - eight-item questionnaire assessing sleep behaviors on a scale of 0 to 3. Higher scores = increased average sleep propensity in daily life
Changes in Emotional Regulation as measured via ERQ | Monthly from baseline through study completion at 8 weeks
  Participants' ability to regulate their emotions appropriately will be quantified via the previously validated Emotional Regulation Questionnaire (ERQ), in which participants will indicate how much they agree with each statement (1, strongly disagree; 7, strongly agree).
Changes in Perceived Stress as measured via PSS | Weekly from baseline through study completion at 8 weeks
  Participants' perceived stress will be quantified via the previously validated Perceived Stress Scale (PSS), which asks participants to report on the frequency of various experiences (0, never; 4, very often) and final scoring suggests lower scores to be associated with lower levels of stress.
Changes in Subjective Sleep as measured via PSQI | Monthly from baseline through study completion at 8 weeks
  Participant's subjective reports of sleep quality will be quantified through the previously validated Pittsburgh Sleep Quality Index (PSQI). Questions are scored into multiple components to determine sleep difficulty in various areas, where higher scores are indicative of greater sleep difficulties; these scores will be compared across timepoints.
Changes in Subjective Anxiety as measured via the STAI | Monthly from baseline through study completion at 8 weeks
  Participants will complete the previously validated State Trait Anxiety Index (STAI) as a measure of subjective anxiety, where higher scores are suggestive of greater anxiety.
Changes in Sleep Disturbances as measured via the Sleep Disorders Questionnaire | Monthly from baseline through study completion at 8 weeks
  Participants will complete a 34 item checklist that has been previously used for screening of a potential sleep disorder; the more items that the participant feels applies to them, the higher the likelihood of the individual having a sleep disorder.
Subjective Success of Commercial Device measured via Questionnaire | Once at the end of week 8
  Following completion of the study, a custom questionnaire will record how successful the participant believes their assigned device was for improving their sleep and well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Rockefeller Neuroscience Institute at West Virginia University, Morgantown, West Virginia, United States